CLINICAL TRIAL: NCT01221233
Title: Lumbar Stabilization Exercises and Neuromuscular Electrical Stimulation: An Investigation of Muscle Size and Function in Older Adults With Chronic Low Back Pain
Brief Title: Investigation of Trunk Muscle Size and Function in Older Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Jaclyn Sions, Assistant Professor, Physical Therapy, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UD005
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES AND Stabilization Exercises (Experimental): Neuromuscular Electrical Stimulation and Lumbar Stabilization Exercises
  Interventions: Other: Neuromuscular Electrical Stimulation
- Moist Heat AND Stabilization Exercises (Active Comparator): Moist Heat and Lumbar Stabilization Exercises
  Interventions: Other: Moist Heat

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation (NMES) to the low back muscles (i.e. spinal extensors) will be applied at the parameters previously used in the knee muscles at the maximal tolerable intensity, which results in a full, sustained isometric contraction of the back muscles. Pad placement will be just below the waist line, with 2, 2X2 inch pads, on either side of the spine. Participants will be positioned on their belly with 2 pillows under their stomach to level the spine and secured to a table using a belt that crosses the buttock.
  The lumbar stabilization program will include exercises targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees).
  Other Names: Lumbar Stabilization Exercises
  Arms: NMES AND Stabilization Exercises
Other: Moist Heat — For participants who do not receive NMES, moist heat will be applied for 15 minutes in a position of comfort for the participant.
  The lumbar stabilization program will include exercises targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees).
  Other Names: Lumbar Stabilization Exercises
  Arms: Moist Heat AND Stabilization Exercises

SUMMARY:
Rehabilitative Ultrasound Imaging (US) is a procedure used to evaluate skeletal muscle size and function to inform clinical practice. US has been shown to be a reliable and valid tool for measuring changes in trunk muscle (i.e. abdominal and back muscle) size and activity during sub-maximal contractions in younger populations. Younger adults with low back pain as compared with healthy adults without pain demonstrate smaller back muscle size, lower back muscle activity, and greater back muscle asymmetry (differences in right side compared with left side).

No trials are published evaluating muscle adaptations using US in response to clinical treatments for low back pain in the older adult population. Increased muscle size and improved muscle symmetry have been reported in younger adults with low back pain who participate in low back stabilization exercises. These exercises use voluntary contractions of the back muscles with prolonged hold times and low loads. Neuromuscular Electrical Stimulation (NMES) is a treatment modality that increases muscle activity when voluntary activity is impaired and increases muscle size. Most studies assessing muscle size and activity in response to NMES have been conducted in the knee muscles (i.e. the quadriceps), while the impact of NMES on the back muscles remains relatively unexplored. Given the potential to evaluate back muscle size and activity with US, this assessment tool may be used to document muscle adaptations to a clinical intervention in older adults with low back pain.

The purpose of this study is to conduct a 6-week clinical trial to determine if NMES plus lumbar stabilization exercises (i.e. NMES AND Stabilization Exercises) is superior to lumbar stabilization exercises (i.e. Moist Heat AND Stabilization Exercises) for improving back muscle size, activity, and side-to-side (i.e. right side versus left side) symmetry in older adults with chronic low back pain (i.e. low back pain of greater than 3 months). Muscle size, activity, and symmetry will be assessed using US before and after the treatments to determine if the treatments positively impact muscle. Secondary clinical measures of success will include improvements in physical, psychological, and social function pre- to post-treatment.

ELIGIBILITY:
Inclusion Criteria: This study will use a sample consisting of 36, English-speaking and English-reading, older male and female adults (ages 60-85 years) with chronic low back pain, i.e. pain of greater than 3 months duration. During the examination, potential participants must have 2/4 of the following for inclusion, based on previous work by Hicks et al, which outlined clinical predictors of success with a trunk muscle stabilization exercise program:

1. Fear-Avoidance Beliefs Questionnaire (FABQ) Physical Activity Sub-Scale score ≥9: The FABQ is a measure of an individual's beliefs regarding the impact of physical activity and work on his/her low back pain. The FABQ is comprised of two sub-scales: physical activity and work. Higher FABQ scores have been shown to predict pain and disability in individuals with chronic low back pain.
2. Aberrant Movement: Aberrant movement may be classified as any one of the following: (1) an "instability catch", defined as deviation from the plane of movement during flexion or extension; (2) "thigh climbing", which is defined as using the hands and pushing on the thighs to assist in obtaining an upright trunk position; (3) a "painful arc of motion", when flexing or returning to upright from a flexed spinal position; or (4) "reversal of the lumbopelvic rhythm", where the trunk is first extended and then the hips and pelvis extend to bring the body upright from a flexed position.
3. Posterior-to-Anterior Segmental Hypermobility: The participant will lie on his/her stomach and the examiner will apply a posterior-to-anterior (back-to-front) force over the spinous processes from S1 to T12 (just below the belt-line to the rib cage). The available mobility will be graded hypermobile (too much motion), normal, or hypomobile (too little motion).
4. Positive Prone Instability Test: The participant will lie on his/her stomach with the legs off the edge of the table and the feet resting on the floor. The examiner will apply a posterior-to-anterior pressure at each spinous process (T12-S1). Any provocation of pain will require the participant to lift their legs off the floor while the pressure is reapplied to the painful level. If the pain subsides with elevation of the legs, this is considered a positive test.

Exclusion Criteria: Exclusion criteria for participants includes (1) history of low back surgery; (2) recent trauma (i.e. motor vehicle accident, fall, etc. ); (3) receipt of services for low back pain within the last 6 months; (4) non-ambulatory or severely impaired mobility (i.e. use of an assistive device greater than a cane); (5) severe hearing or visual impairment; (6) non-mechanical low back pain; (7) neurological disorder; (8) presence of an acute illness; (9) diagnosis of scoliosis; (10) symptoms related to the back below the knee; (11) presence of a pacemaker; (12) participation in R21 clinical trial ongoing at the University of Delaware Physical Therapy Clinic; or (13) the inability to participate in the study for the full six weeks for any known reason (i.e. moving away, extended vacation). Potential participants will also be excluded if during the evaluation any of the following are found:

1. score < 24 on the Folstein Mini-Mental State Examination (MMSE): As scores greater than or equal to 24 may identify individuals who are cognitively intact, this screening tool will exclude those older adults with questionable reliability (i.e. consistency) on the self-report questionnaires secondary to cognitive impairment.
2. Modified Oswestry Low Back Pain Questionnaire (mOSW) score < 14 percent: This questionnaire will exclude those individuals with chronic low back pain who demonstrate minimal low back pain-related disability. Individuals with minimal disability may not be representative of those seeking outpatient physical therapy services for their back pain.
3. Facial Pain Scale-Revised (FPS-R) "worst" low back pain rating in last 24 hours of < 3/10: Pain rating ≥ 3/10 is being used in the hopes of recruiting a group of individuals who may be representative of those likely to seek clinical services for their low back pain. Also, all FPS-Rs ("current", "best", and "worst") will be used to document the impact of treatment on self-reported pain.
4. Inability to tolerate lying on belly with legs straight: This is a requirement for our standardized position for ultrasound.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-02-14 (Actual); Primary Completion 2011-11-22 (Actual); Study Completion 2011-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NMES AND Stabilization Exercises: Neuromuscular Electrical Stimulation and Lumbar Stabilization Exercises
  Neuromuscular Electrical Stimulation: Neuromuscular Electrical Stimulation (NMES) to the low back muscles (i.e. spinal extensors) will be applied at the parameters previously used in the knee muscles at the maximal tolerable intensity, which results in a full, sustained isometric contraction of the back muscles. Pad placement will be just below the waist line, with 2, 2X2 inch pads, on either side of the spine. Participants will be positioned on their belly with 2 pillows under their stomach to level the spine and secured to a table using a belt that crosses the buttock.
  The lumbar stabilization program will include exercises targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees).
- Moist Heat AND Stabilization Exercises: Moist Heat and Lumbar Stabilization Exercises
  Moist Heat: For participants who do not receive NMES, moist heat will be applied for 15 minutes in a position of comfort for the participant.
  The lumbar stabilization program will include exercises targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees).
Period: Overall Study
Arm/Group | NMES AND Stabilization Exercises | Moist Heat AND Stabilization Exercises
Started | 18 | 20
Completed | 15 | 19
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES AND Stabilization Exercises | Moist Heat AND Stabilization Exercises | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (7.6) | 71.3 (7.7) | 71.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 8 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 17 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 19 | 34
Modified Oswestry Disability Index [Mean (Standard Deviation); unit: %] — A self-report questionnaire evaluating low back pain-related disability, where higher scores indicate greater disability.
  The total score is reported from 0-100%.
  % | 25.5 (8.7) | 22.2 (7.9) | 23.6 (8.3)
Fear-Avoidance Beliefs Questionnaire-Physical Activity Subscale [Mean (Standard Deviation); unit: scores on a scale] — A self-report questionnaire evaluating fear-related to physical activity, where higher scores are indicative of greater fear that activity may make back pain worse.
  Physical activity subscale scores range from 0-24.
  scores on a scale | 13.7 (4.4) | 15.2 (6.5) | 14.5 (5.7)
Left L4/5 Lumbar Multifidus Activity [Mean (Standard Deviation); unit: percentage of activity] — Lumbar multifidus activity is obtained from ultrasound imaging using brightness-mode, where two images, resting and contracted are obtained side-by-side. Measurements are obtained from the facet joint to the last pixel before the muscle's fascial line. Measurements are used in the following calculation to determine muscle activity: (contracted thickness-resting thickness)/resting thickness. Results are reported for the average of 3 sets of images as a percentage, where higher percentages indicate greater muscle activity. Percentages may range from 0% (i.e. no activity) to 100%.
  percentage of activity | 11.1 (5.6) | 12.3 (4.9) | 11.8 (5.2)
Right L4/5 Lumbar Multifidus Activity [Mean (Standard Deviation); unit: percentage of activity] — Lumbar multifidus activity is obtained from ultrasound imaging using brightness-mode, where two images, resting and contracted are obtained side-by-side. Measurements are obtained from the facet joint to the last pixel before the muscle's fascial line. Measurements are used in the following calculation to determine muscle activity: (contracted thickness-resting thickness)/resting thickness. Results are reported for the average of 3 sets of images as a percentage, where higher percentages indicate greater muscle activity. Percentages may range from 0% (i.e. no activity) to 100%.
  percentage of activity | 9.5 (6.0) | 11.8 (4.4) | 10.8 (5.3)
Left L4 Paraspinal Muscle Size [Mean (Standard Deviation); unit: cm2] — Paraspinal muscle size is obtained from ultrasound imaging using brightness-mode, where the multifidus and longissimus are imaged just adjacent to the spinous process. Cross-sectional measurements are obtained by tracing just insides the muscle fascial lines. Measurements from 3 separate images were averaged. Greater sizes are generally better. Muscle size varies by vertebral level and by other factors, such as sex and body mass. Typical values have not been reported for this age-group.
  cm2 | 11.6 (2.0) | 12.0 (2.0) | 11.9 (2.0)
Right L4 Paraspinal Muscle Size [Mean (Standard Deviation); unit: cm2] — Paraspinal muscle size is obtained from ultrasound imaging using brightness-mode, where the multifidus and longissimus are imaged just adjacent to the spinous process. Cross-sectional measurements are obtained by tracing just insides the muscle fascial lines. Measurements from 3 separate images were averaged. Greater sizes are generally better. Muscle size varies by vertebral level and by other factors, such as sex and body mass. Typical values have not been reported for this age-group.
  cm2 | 11.1 (2.1) | 11.4 (1.8) | 11.2 (1.9)
L4 Paraspinal Cross-Sectional Area Asymmetry [Mean (Standard Deviation); unit: percent asymmetry] — Paraspinal muscle size is obtained from ultrasound imaging using brightness-mode, where the multifidus and longissimus are imaged just adjacent to the spinous process. Cross-sectional measurements are obtained by tracing just insides the muscle fascial lines. Side-to-side asymmetry was calculated as percent side-to-side difference = [(largest value/smallest value)*100]-100), so 0% indicates right and left paraspinal muscles are equal. Typical cross-sectional area asymmetry in this age group is unknown, but theoretically greater symmetry (i.e. lower percentages) would be ideal.
  percent asymmetry | 14.0 (13.3) | 10.1 (7.8) | 11.8 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Percent Change From Baseline in L4 Paraspinal Cross-Sectional Area Asymmetry at 6 Weeks Between Intervention Arms
Description: Percent change (baseline-6 weeks)/baseline X100% was calculated for each participant in each intervention arm and then these differences were compared using a Mann-Whitney U test since data did not meet parametric assumptions.
Time Frame: Baseline and 6 Weeks
Population: Analyses were only completed on participants who completed the randomized clinical trial.
Measure: Median (Inter-Quartile Range); unit: % change
Groups:
- NMES AND Stabilization Exercises: Neuromuscular Electrical Stimulation (NMES) and Lumbar Stabilization Exercises
  Participants received a physical therapy intervention 2 times per week for 6 weeks that consisted of a lumbar stabilization exercise program targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees) followed by NMES set to portable 300PV unit by EMPI (St. Paul, MN) was set to the following: 50 bursts per second, 12 seconds of contraction, 50 seconds of rest, a 2 second ramp, 400 microseconds, and a treatment time of 20 minutes
- Moist Heat AND Stabilization Exercises: Participants received a physical therapy intervention 2 times per week for 6 weeks that consisted of a lumbar stabilization exercise program targeting the back muscles in three positions: standing, prone (belly), and quadruped (hands and knees) followed by 20 minutes of moist heat to the low back region.
Arm/Group | NMES AND Stabilization Exercises | Moist Heat AND Stabilization Exercises
Number analyzed (Participants) | 15 | 19
% change | 0 [-57.1 to 104.3] | -17.6 [-51.1 to 250.0]
Statistical Analysis 1: Comparison: NMES AND Stabilization Exercises; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 17.6

ADVERSE EVENTS:
Time Frame: Baseline, 6 weeks of intervention, and 6-week follow-up.
Description: Adverse events were reported by study personnel in accordance with the University of Delaware Institutional Review Board for Human Subjects Research. Adverse event definitions as described in the Common Terminology Criteria for Adverse Events (CTCAE) from the National Institutes of Health are used for reporting.
Groups:
- NMES AND Stabilization Exercises: Neuromuscular Electrical Stimulation (NMES) and Lumbar Stabilization Exercises
Arm/Group | NMES AND Stabilization Exercises | Moist Heat AND Stabilization Exercises
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 1/18 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NMES AND Stabilization Exercises (N=18) | Moist Heat AND Stabilization Exercises (N=20)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lack of long-term follow-up; short-duration intervention may have been insufficient for muscle change

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT01221233/Prot_SAP_000.pdf